CLINICAL TRIAL: NCT03222453
Title: The Third Affiliated Hospital of Guangzhou Medical University
Brief Title: Thalassemia Treatment Based on the Stem Cell Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xiaofang Sun (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Guangzhou Institutes of Biomedicine and Health Chinese Academy of Sciences (Unknown); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Xiaofang Sun, Principal Investigator, The Third Affiliated Hospital of Guangzhou Medical University
Organization: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201508020258
Record Dates: First submitted 2017-06-23; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Beta-Thalassemia
Keywords: thalassemia; stem cell
MeSH Terms: conditions — beta-Thalassemia; Thalassemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Patient (Experimental): Hematopoetic stem cells differentiated from beta-thalassemia induced pluripotent stem cells.
  Interventions: Biological: Hematopoetic stem cells
- non-intervention Patient (No Intervention): No treatment

INTERVENTIONS:
Biological: Hematopoetic stem cells — Patient will inject with hematopoetic stem cells differentiated from beta-thalassemia induced pluripotent stem cells
  Arms: Intervention Patient

SUMMARY:
In order to study the transplantation effect of hematopoetic stem cells from beta-thalassemia induced pluripotent stem cells. We applied clinical grade source of autologous hematopoietic stem cell for the treatment of beta-thalassemia patients, detecting the homing of hematopoietic stem cell transplantation, the differentiation of hematopoietic stem cells in vivo and the hemoglobin beta-chain (HBB) protein expression in the body of recovery, etc., as well as to make a research on the efficacy and safety of hematopoietic stem cells from beta-thalassemia induced pluripotent stem cells.

DETAILED DESCRIPTION:
1. On a Good Manufacturing Practice(GMP) condition, we establish non-exotic of different mutation types of beta-thalassemia -induced pluripotent stem cells（iPS） and make a comparisons of the stability and the differentiation of efficiency of these iPS cells inducing from different sources with foreign gene integration.
2. Using the technique of artificial nuclease and in situ repairmen, we establish efficient system for different beta-thalassemia mutation site and in view of the security of these system.
3. Establish a repaired beta-thalasemia gene mutated differentiation of iPS technology system.
4. Build a functional gene therapy self-limiting slow viruses, optimizing the preparation system and to establish a virus preparation of infection of hematopoietic stem cell technology system under the GMP condition.
5. Establish humanized beta-mice model, evaluate the safety of the iPS cell of gene therapy and efficiency before the clinical experiment.
6. Improve the existing hematopoietic stem cell transplant(HSCT) clinical application solutions, detect rate of graft rejection, rate of transplantation and other indicators, finish the evaluation of application by clinical cases.

ELIGIBILITY:
Inclusion Criteria:

1. The genetic diagnosis confirmed homozygous for beta to poverty or double heterozygote, clinical severe anemia;
2. Aged 1 ~ 18 years old, no obvious iron overload cause organ damage;
3. Has a suitable donor HLA high resolution;
4. The informed consent

Exclusion Criteria:

1. There has been a significant increase in the level of tumor markers (AFP/CEA/CA199 / CA125) in the past five years.
2. Serious primary diseases such as cardiovascular, liver and hematopoietic systems; Those who have major organs with serious function; An adrenal disease or other disease that causes the organ failure of the organ;
3. An autoimmune disease, a family history of genetic disease, and an abnormal thyroid function;
4. Peripheral blood chromosome checking for nuclear aliens;
5. HIV, hepatitis b or hepatitis c;
6. A person with a history of severe drug allergies or an allergic person;
7. Those who do not expect to live for more than one year;
8. The researchers suggest that the patient may have a potential or have a disorder (such as an uncontrolled infection, right heart failure, pulmonary hypertension) that is interfering with this study.
9. In the first six months, alcohol and other substance abuse were not allowed;
10. Subjects who participated in other clinical trials or participated in other clinical trials within 3 months.

Ages: 1 Year to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Clinical diagnosis.
Enrollment: 2 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
The check of granulocyte transplantation-granulocyte plant living standards | 3 days
  Granulocyte plant living standards for three days in a row after transplantation granulocyte should be greater than 0.5 x 109 / L,
The check of granulocyte transplantation-platelet plant living standards | seven consecutive days
  Platelet plant living standard for seven consecutive days after transplantation the platelet should be greater than 20 x 109 / L and infusion.
Effect of cell transplantation | seven days
  The granulocyte plant living standards and platelet plant living standards will be combined to measure the effect of cell transplantation.

IPD SHARING:
Plan to Share IPD: Undecided